CLINICAL TRIAL: NCT05420077
Title: Phase 1, Open-Label, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Immunogenicity of RVM-V001 in Healthy Individuals Aged 18-65 Years Previously Vaccinated With BNT162b2 and mRNA-1273
Brief Title: Safety and Immunogenicity of RVM-V001 in Healthy Individuals Previously Vaccinated With BNT162b2 and mRNA-1273
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The landscape of the study area changed, making it impossible to continue the study.
Sponsor: RVAC Medicines (US), Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: RV002
Record Dates: First submitted 2022-06-07; First posted 2022-06-15 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Infectious Disease; COVID-19
MeSH Terms: conditions — Communicable Diseases; COVID-19 | interventions — RVM-V001 COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RVM-V001 10 µg (Experimental): RVM-V001-10 µg administered as a single dose of by intramuscular injection on Day 1
  Interventions: Biological: RVM-V001 10 µg
- RVM-V001 30 µg (Experimental): RVM-V001-30 µg administered as a single dose of by intramuscular injection on Day 1
  Interventions: Biological: RVM-V001 30 µg
- RVM-V001 60 µg (Experimental): RVM-V001-60 µg administered as a single dose of by intramuscular injection on Day 1
  Interventions: Biological: RVM-V001 60 µg

INTERVENTIONS:
Biological: RVM-V001 10 µg — Low Dose
  Arms: RVM-V001 10 µg
Biological: RVM-V001 30 µg — Mid Dose
  Arms: RVM-V001 30 µg
Biological: RVM-V001 60 µg — High Dose
  Arms: RVM-V001 60 µg

SUMMARY:
Phase 1, open-label, dose-escalation study to evaluate the safety, tolerability, and immunogenicity of RVM-V001 administered as a single intramuscular injection in healthy adults. Three dose levels will be evaluated, with progression from low- to high-dose level based on the assessment of safety and tolerability. The study will be conducted at one or more sites in Australia.

DETAILED DESCRIPTION:
Approximately 54 healthy non-pregnant female and male adults aged 18-65 years inclusive are planned to be enrolled in the study. All subjects will have completed either a 2-dose primary vaccination series with Pfizer Biontech-BNT162b2 SARS-CoV-2 vaccine (P) or Moderna mRNA-1273 (M) (as authorized/approved or as investigational product in a clinical trial), OR have completed the primary series and one homologous booster of Pfizer Biontech-BNT162b2 or mRNA-1273 i.e, P-P-P and M-M-M; the last dose in all cases should have been administered at least 6 months prior to enrollment.

This study is composed of 3 dose groups, Groups 1, 2 and 3 per dose level. 18 eligible subjects in each dose group will receive RVM-V001 on Study Day 1 via intramuscular (IM) injection into deltoid muscle of the non-dominant arm.

Subjects will be sequentially assigned to a dose group beginning with Group 1 (10 µg RVM-V001) based on the timing of completion of screening. As a precautionary step, 3 sentinel subjects, at least one male and one female will be used within each dose group. Enrollment of each dose group will start with the 3 sentinel subjects. After at least 2 days from the time of study vaccine administration of the 3 sentinel subjects, the 2-day safety data will be collected and reviewed by the principal investigator and local medical monitor. Should there be no safety concerns, the remaining subjects in the same dose group can be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Male and female healthy volunteers.
* Is age 18 and 65 years inclusive on Study Day 1.
* Judged by the investigator to be healthy based on medical history, physical examination, vital signs, and no significant electrocardiogram (ECG) abnormalities performed at screening.
* Able to provide informed consent form.
* Able and willing to comply with all study procedures over follow-up period of approximately 6 months.
* Have completed either a 2-dose primary vaccination series with Pfizer Biontech-BNT162b2 SARS-CoV-2 vaccine (P) or Moderna mRNA-1273 (M) (as authorized/approved or as investigational product in a clinical trial), OR have completed the primary series and one homologous booster of Pfizer Biontech-BNT162b2 or mRNA-1273 i.e, P-P-P and M-M-M; the last dose in all cases should have been administered at least 6 months prior to enrollment.
* Body mass index of 18-32 kg/m2, inclusive, at screening.
* For female subjects with childbearing potential: must agree to avoid pregnancy from 21 days prior to Study Day 1 until at least 90 days after last study vaccination. Women physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses if menopausal) in sexual relationships with men must use an acceptable method of avoiding pregnancy during this period. Acceptable methods of avoiding pregnancy include a sterile sexual partner, hormonal contraceptives (oral, injection, transdermal patch, or implant), vaginal ring, intrauterine device (IUD), or the combination of a condom or diaphragm.
* Men must be willing to refrain from sperm donation, starting after screening until 90 days after receiving the last vaccination.
* Male and female subjects must use a barrier method of contraception, from 21 days prior to Study Day 1 until at least 90 days after last study vaccination. Barrier methods of contraception include:

  * Male condoms
  * Female condoms
  * Female diaphragm ('cap')

Exclusion Criteria:

* Documented history of COVID-19 within 6 months prior to enrollment.
* Positive reverse transcription - polymerase chain reaction (RT-PCR) test for SARS-CoV-2 within 2 days of screening
* Received any COVID-19 vaccine other than BNT162b2 or mRNA-1273.
* Received more than 3 doses of any mRNA COVID-19 vaccine.
* Pregnant or breastfeeding or intending to become pregnant or father children within the projected duration of the trial.
* Currently working in an occupation with a high risk of exposure to SARS-CoV-2 (eg, Healthcare worker, emergency response personnel having direct interactions with or providing direct care to patients).
* History of infection of Middle East respiratory syndrome (MERS), or Severe Acute respiratory syndrome (SARS).
* Positive serology test results for hepatitis C virus antibody, HIV antibody, hepatitis B virus surface antigen at Screening.
* Currently taking marketed, investigational, off-label product for the prevention of MERS, SARS, or COVID-19.
* Is currently participating in or has participated in a study with an investigational product within 30 days preceding Day 1.
* Fever (tympanic temperature > 37.5 degree C), dry cough, fatigue, nasal obstruction, runny nose, sore throat, myalgia, diarrhea, shortness of breath or dyspnea within 14 days before administration
* Abnormal indicators, such as blood biochemistry, blood routine and urine routine deemed clinically significant by the investigator, or the value is beyond Grade 1 per toxicity grading scale.
* History of severe allergic reactions (such as acute anaphylaxis, urticaria, skin eczema, dyspnea, angioneurotic edema or abdominal pain) or allergy to known composition of RVM-V001 vaccine.
* History of convulsion, epilepsy, encephalopathy or severe mental illness.
* Diagnosed with congenital malformations or developmental disorders, genetic defects, severe malnutrition.
* Diagnosed with severe liver and kidney diseases, uncontrollable hypertension (systolic pressure >140 mmHg, diastolic pressure >90 mmHg), diabetic complications, malignant tumors, acute viral or bacterial infections or acute onset of chronic disease.
* Diagnosed with congenital or acquired immune deficiency, HIV infection, lymphoma, leukemia or other autoimmune diseases
* History of coagulation dysfunction (eg, Coagulation factor deficiency, coagulation disease).
* Vaccinated with live attenuated vaccine within 1 month, or other vaccine within 14 days before vaccination.
* Receiving immunotherapy or inhibitor therapy within 3 months (consistently oral or infusion for more than 14 days).
* Received systemic immunosuppressants within 4 months prior to vaccination or anticipating the need for immunosuppressant at any time during participation in the study. Topical or inhaled treatment is allowed if not used within 14 days prior to vaccination.
* Receiving blood products within 3 months before administration
* History of alcohol or drug abuse within 3 years before first vaccination.
* Has donated 450ml or greater of blood within 28 days prior to vaccination.
* History of anaphylaxis or angioedema including but not limited to history of anaphylaxis after any vaccine.
* Any condition that, in the opinion of the investigator, would pose a health risk to the subject if enrolled or could interfere with evaluation of the study vaccine or has interpretation of study results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Number of subjects with solicited adverse events | Day 1 to Day 8 post dose
Number of subjects with solicited systemic adverse events | Day 1 to Day 8 post dose
Number of subjects with unsolicited adverse events | Day 1 to Day 29 post dose
Number of subjects with SAEs, SUSARs, MAAEs and AESIs | Day 1 to Day 180 post dose
Changes in safety laboratory parameters from baseline by the Food and Drug Administration (FDA) toxicity grading scale. | Day 1 to Day 180 post dose
GMT of of neutralizing antibody (pseudoviral neutralization assay) against Wuhan strain | Baseline and Day 29
GMT of neutralizing antibody (pseudoviral neutralization assay) against Omicron and Delta variants of SARS-CoV-2 | Baseline and Day 29
GMT of serum binding antibodies (IgG) by ELISA | Baseline and Day 29
Seroresponse rate for neutralizing antibody | Day 29
  SRR percentage of subjects with ≥4-fold increase of antibody titer over baseline
Seroresponse rate for binding antibodies (IgG) by ELISA | Day 29
  SRR percentage of subjects with ≥4-fold increase of antibody titer over baseline
Geometric Mean Fold Rise (GMFR) of SARS-CoV-2 Neutralizing Antibody | Day 29
Geometric Mean Fold Rise (GMFR) of binding antibodies (IgG) by ELISA | Day 29

SECONDARY OUTCOMES:
GMT of of neutralizing antibody (pseudoviral neutralization assay) against Wuhan strain | Days 15 and 180
GMT of neutralizing antibody (pseudoviral neutralization assay) against Omicron and Delta variants of SARS-CoV-2 | Days 15 and 180
GMT of serum binding antibodies (IgG) by ELISA | Days 15 and 180
Seroresponse rate for neutralizing antibody | Days 15 and 180
  SRR percentage of subjects with ≥4-fold increase of antibody titer over baseline
Seroresponse rate for binding antibodies (IgG) by ELISA | Days 15 and 180
  SRR percentage of subjects with ≥4-fold increase of antibody titer over baseline
Geometric Mean Fold Rise (GMFR) of SARS-CoV-2 Neutralizing Antibody | Days 15 and 180
Geometric Mean Fold Rise (GMFR) of binding antibodies (IgG) by ELISA | Days 15 and 180

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Northern Beaches Clinical Research, Brookvale, New South Wales
  - Core Research Group Pty Ltd, Brisbane, Queensland